CLINICAL TRIAL: NCT05043129
Title: Safety and Immune Response of COVID-19 Vaccination in Patients With HIV Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Hong Ren, Dr/ Prof., The Second Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2021-43
Record Dates: First submitted 2021-09-10; First posted 2021-09-14 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: HIV Infections; Covid19
MeSH Terms: conditions — HIV Infections; COVID-19 | interventions — Biological Products; COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV infenction/AIDS: experimental group
  Interventions: Biological: Biological/Vaccine: SARS-COV-2 VACCINE
- Healthy population: Control group
  Interventions: Biological: Biological/Vaccine: SARS-COV-2 VACCINE

INTERVENTIONS:
Biological: Biological/Vaccine: SARS-COV-2 VACCINE — The antibody titer and adverse reactions were observed.

SUMMARY:
On 11 February 2020, the International Committee for the Classification of Viruses named the disease caused by SAＲS-CoV-2 infection in humans as the new coronavirus pneumonia (coronavirus disease 2019, COVID-19). People infected with human immunodeficiency virus (HIV) are affected by their underlying diseases and are listed by the World Health Organization (WHO) as a high-risk population of SARS-CoV-2 infection.To evaluate the safety and effectiveness of COVID-19 vaccine in those patients with human immunodeficiency virus infection , and to guide the COVID-19 vaccination more scientifically, reasonably and effectively, this study was carried out.

DETAILED DESCRIPTION:
People infected with human immunodeficiency virus (HIV), affected by their underlying diseases, are listed by the World Health Organization (WHO) as a high-risk population for SARS-CoV-2 infection.. More attention should be paid to personal protection and disease prevention. Vaccination of COVID-19 can effectively prevent COVID-19 virus infection and delay or prevent patients from developing into critical illness and reduce mortality. The safety and effectiveness of COVID-19 vaccine in this population were evaluated in order to play a scientific and theoretical supporting role in guiding COVID-19 vaccination more scientifically, reasonably and effectively. The samples of this study were collected and tested in the second affiliated Hospital of Chongqing Medical University. Patients with contraindications for vaccination will be excluded. The detected indexes included blood routine test, CD4, HIV virus load, COVID-19 antibody titer, antibody duration and other indexes of healthy people (control group) and HIV infenction people after vaccination ( 1, 3, 6 months after vaccination). The adverse reactions related to the vaccine were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. HIV infection group: a. The HIV positive diagnosis is clear; b. 18-80 years old; c. Has been vaccinated against the COVID-19 ; d. Volunteer to participate in the project;
2. Healthy control group: a. HIV negative; b. Age 18-80 years old; c. The COVID-19 vaccination has been completed; d. Volunteer to participate in the project

Exclusion Criteria:

1. Previous confirmed case of COVID-19
2. confirmed contact history of COVID-19
3. vaccination contraindications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV infected persons vaccinated with COVID-19 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-04 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events after injection | 1 month after vaccination
  The vaccine-related adverse reactions (such as fever, dizziness, fatigue, myalgia, etc.) were recorded and its safety was evaluated.
Number of participants with adverse events after injection | 3 months after vaccination
  The vaccine-related adverse reactions (such as fever, dizziness, fatigue, myalgia, etc.) were recorded and its safety was evaluated.
Number of participants with adverse events after injection | 6 months after vaccination
  The vaccine-related adverse reactions (such as fever, dizziness, fatigue, myalgia, etc.) were recorded and its safety was evaluated.

SECONDARY OUTCOMES:
Titer and duration of COVID-19 antibody production after vaccination | 1 month after vaccination
  The titer and duration of COVID-19 antibody were produced at 1 month
Titer and duration of COVID-19 antibody production after vaccination | 3 months after vaccination
  The titer and duration of COVID-19 antibody were produced at 3 months
Titer and duration of COVID-19 antibody production after vaccination | 6 months after vaccination
  The titer and duration of COVID-19 antibody were produced at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hong Ren, PHD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- China, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu Z, Shi L, Wang Y, Zhang J, Huang L, Zhang C, Liu S, Zhao P, Liu H, Zhu L, Tai Y, Bai C, Gao T, Song J, Xia P, Dong J, Zhao J, Wang FS. Pathological findings of COVID-19 associated with acute respiratory distress syndrome. Lancet Respir Med. 2020 Apr;8(4):420-422. doi: 10.1016/S2213-2600(20)30076-X. Epub 2020 Feb 18. No abstract available. PMID 32085846
- [Background] Zhu FC, Guan XH, Li YH, Huang JY, Jiang T, Hou LH, Li JX, Yang BF, Wang L, Wang WJ, Wu SP, Wang Z, Wu XH, Xu JJ, Zhang Z, Jia SY, Wang BS, Hu Y, Liu JJ, Zhang J, Qian XA, Li Q, Pan HX, Jiang HD, Deng P, Gou JB, Wang XW, Wang XH, Chen W. Immunogenicity and safety of a recombinant adenovirus type-5-vectored COVID-19 vaccine in healthy adults aged 18 years or older: a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2020 Aug 15;396(10249):479-488. doi: 10.1016/S0140-6736(20)31605-6. Epub 2020 Jul 20. PMID 32702299
- [Background] Madhi SA, Baillie V, Cutland CL, Voysey M, Koen AL, Fairlie L, Padayachee SD, Dheda K, Barnabas SL, Bhorat QE, Briner C, Kwatra G, Ahmed K, Aley P, Bhikha S, Bhiman JN, Bhorat AE, du Plessis J, Esmail A, Groenewald M, Horne E, Hwa SH, Jose A, Lambe T, Laubscher M, Malahleha M, Masenya M, Masilela M, McKenzie S, Molapo K, Moultrie A, Oelofse S, Patel F, Pillay S, Rhead S, Rodel H, Rossouw L, Taoushanis C, Tegally H, Thombrayil A, van Eck S, Wibmer CK, Durham NM, Kelly EJ, Villafana TL, Gilbert S, Pollard AJ, de Oliveira T, Moore PL, Sigal A, Izu A; NGS-SA Group; Wits-VIDA COVID Group. Efficacy of the ChAdOx1 nCoV-19 Covid-19 Vaccine against the B.1.351 Variant. N Engl J Med. 2021 May 20;384(20):1885-1898. doi: 10.1056/NEJMoa2102214. Epub 2021 Mar 16. PMID 33725432
- [Background] Haynes BF. SARS-CoV-2 and HIV-1 - a tale of two vaccines. Nat Rev Immunol. 2021 Sep;21(9):543-544. doi: 10.1038/s41577-021-00589-w. Epub 2021 Jul 16. PMID 34272508
- [Background] Treskova-Schwarzbach M, Haas L, Reda S, Pilic A, Borodova A, Karimi K, Koch J, Nygren T, Scholz S, Schonfeld V, Vygen-Bonnet S, Wichmann O, Harder T. Pre-existing health conditions and severe COVID-19 outcomes: an umbrella review approach and meta-analysis of global evidence. BMC Med. 2021 Aug 27;19(1):212. doi: 10.1186/s12916-021-02058-6. PMID 34446016
- [Derived] Ao L, Lu T, Cao Y, Chen Z, Wang Y, Li Z, Ren X, Xu P, Peng M, Chen M, Zhang G, Xiang D, Cai D, Hu P, Shi X, Zhang D, Ren H. Safety and immunogenicity of inactivated SARS-CoV-2 vaccines in people living with HIV. Emerg Microbes Infect. 2022 Dec;11(1):1126-1134. doi: 10.1080/22221751.2022.2059401. PMID 35369854